CLINICAL TRIAL: NCT06557031
Title: Clinical Performance Study of the ABTest Card® Device.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diagast (Industry)
Collaborators: Soladis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPSP_23-03
Record Dates: First submitted 2024-08-07; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Transfusion Reaction
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Intervention Model Description: In situ used for near patient In vitro Medical device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ABTest Card®REF and ABTest Card®NEW — Pre transfusional control with the ABTest Card®REF device (predicate device) and the ABTest Card®NEW device (investigational device).

SUMMARY:
The study aims to confirm the performance equivalence of the in vitro diagnostic device ABTest Card®REF with the ABTest Card®NEW device.

DETAILED DESCRIPTION:
Following some changes in the ABTest Card® raw materials, a new validation of the associated clinical performances is required. Raw materials of the ABTest Card® are : Triton, Cleanis, Tween, Yellow, Blue dye and the blood segment opener device.

According to the regulatory text "Common specifications for certain class D in vitro diagnostic medical devices in accordance with Regulation (EU) 2017/746 of the European Parliament and of the Council", 90% of the results will be derived from the performance study carried out at the DIAGAST laboratory on tube left over and blood bag, and 10% of the results will be derived from the use of the device in a real situation ("at the bedside").

The Regulation 2017/746 (IVDR) on IVDMD, has been effective since May 2022 with transitional periods. The IVDR replaces the current EU Directive (98/79/EC) to ensure a higher level of health and safety for the making available and putting into service of medical devices on the EU market. As the ABTest Card® is already CE marked under Directive 98/79/EC as List IIA product, this study is part of the device's post-marketing performance monitoring.

The purpose of this study is to document and verify the clinical performance of the ABTest Card® device in combination with the new raw materials used for manufacturing (ABTest Card®NEW), by comparing the results obtained with the ABTest Card®REF, already commercialised and used routinely by the study sites.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old for the category marked with *.
* Undergo capillary blood sampling ;
* Belong to one of the clinical categories:
* Patient in need of blood transfusion without any pathology known to have an impact on transfusion act* ;
* Patient in need of blood transfusion suffering from congenital erythrocyte pathology (sickle cell anaemia, beta thalassemia)* ;
* Patient in need of blood transfusion suffering from haematology disease (e.g. cancer), or undergoing haemodialysis* ;
* Patient with cold agglutinin* ;
* Premature patient with gestational age < 37 weeks or newborn ≤27 days old in need of blood transfusion ;
* Newborn eligible for the Guthrie Test ;
* Newborn eligible for the glycaemic test.
* Have health care insurance ;
* Have given his/her written consent (or legal representative in the case of a newborn) ;

Exclusion Criteria:

* Pregnant woman ;
* Person deprived of liberty ;
* Unconscious person ;
* Person under guardianship or trusteeship ;
* For paediatric clinical category: age ≥28 days and <18 years old.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Concordance obtained on patient blood type between ABTest Card®NEW and ABTest Card®REF results. | 1 day.
  Comparison of the "patient" blood type determined from the results of the ABTest Card®NEW device (A, B, AB, O) with the "patient" blood type determined from the results of the ABTest Card®REF device (A, B, AB, O).
  There is concordance if the two "patient" blood types are identical.

SECONDARY OUTCOMES:
Concordance obtained on blood bag blood type between the ABTest Card®NEW and ABTest Card®REF results. | 1 day.
  Comparison of the "donor" blood type determined from the results of the ABTest Card®NEW device (A, B, AB, O) with the "donor" blood type determined from the results of the ABTest Card®REF device (A, B, AB, O).
  There is concordance if the two "donor" blood types are identical.
Concordance obtained between blood type information from medical record and patient results obtained by ABTest Card®REF. | 1 day.
  Comparison of the "patient" blood type determined from the results of the ABTest Card®REF device (A, B, AB, O) with the "patient" blood type in the medical record (A, B, AB, O).
  There is concordance if the two "patient" blood types are identical.
Concordance obtained between blood bag labelling information and blood bag results obtained by ABTest Card®REF. | 1 day.
  Comparison of the "donor" blood type determined from the results of the ABTest Card®REF device (A, B, AB, O) with the "donor" blood type shown on the blood bag label (A, B, AB, O).
  There is concordance if the two "donor" blood types are identical.
Blood compatibility between the blood bag and the patient for the ABTest Card®NEW. | 1 day.
  Comparison of the "patient" blood type determined from the results of the ABTest Card®NEW device (A, B, AB, O) with the "donor" blood type determined from the results of the ABTest Card®NEW device (A, B, AB, O).
  There is blood compatibility if the two blood types follow specific associations.
Blood compatibility between the blood bag and the patient for the ABTest Card®REF. | 1 day.
  Comparison of the "patient" blood type determined from the results of the ABTest Card®REF device (A, B, AB, O) with the "donor" blood type determined from the results of the ABTest Card®REF device (A, B, AB, O).
  There is blood compatibility if the two blood types follow specific associations.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: Undecided